CLINICAL TRIAL: NCT03104426
Title: Randomized Controlled Trial on the Use of EPO to Reduce Top-up Transfusions in Neonates With Red Blood Cell Alloimmunization Treated With Intrauterine Transfusions
Brief Title: EPO-4-Rhesus Study
Acronym: EPO-4-Rhesus
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanquin-LUMC J.J van Rood Center for Clinical Transfusion Research (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P17.102
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Erythroblastosis, Fetal; Erythroblastosis Fetalis, Rh Disease; Erythroblastosis Fetalis Due to RH Antibodies; Erythroblastosis Fetalis Due to Isoimmunization
Keywords: Hemolytic disease of the fetus and newborn; HDFN; Red blood cell alloimmunization
MeSH Terms: conditions — Erythroblastosis, Fetal | interventions — Darbepoetin alfa

STUDY DESIGN:
Intervention Model Description: RCT with unblinded treatment allocation 1:1 ratio. Either treatment with darbepoetin alfa or "standard care". No placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Darbepoetin alfa group (Active Comparator): Group treated with darbepoetin alfa (Aranesp) 10microg/kg once a week for a period of 8 weeks.
  Interventions: Drug: Darbepoetin Alfa
- Control group (No Intervention): "Standard care" which involves close monitoring of hemoglobin levels and if necessary, top-up red cell transfusion.

INTERVENTIONS:
Drug: Darbepoetin Alfa — Darbepoetin alfa dosage 10microg/kg once a week for 8 weeks
  Other Names: Aranesp
  Arms: Darbepoetin alfa group

SUMMARY:
Up to 80% of infants with hemolytic disease due to maternal alloimmunization, treated with IUT, require at least one top-up transfusion for late anemia during the first 3 months of life. Erythropoietin deficiency is also considered as a possible contributing factor to late anemia and therefore we will assess the role of EPO (darbepoetin alfa) in the treatment of these infants.

DETAILED DESCRIPTION:
The mainstay of antenatal treatment of fetal anemia due to red cell alloimmunization is (serial) IUT. The mainstay of postnatal treatment in HDN is (1) intensive phototherapy and exchange transfusion to treat hyperbilirubinemia and prevent kernicterus, and (2) top-up transfusions to treat anemia. Up to 80% of infants with HDN treated with IUT require at least one top-up transfusion for late anemia during the first 3 months of life.

Several risk factors for late anemia have been reported, including serial IUT (due to bone marrow suppression), severity of HDN, reduced use of exchange transfusions during the neonatal period and reduced survival of transfused red blood cells. Finally, erythropoietin deficiency is also considered as a possible contributing factor to late anemia.

EPO has been increasingly used in neonates to prevent or reduce neonatal anemia without short or long-term adverse effects. Several small studies and casuistic reports suggest that neonates with HDN may benefit from treatment with EPO to reduce the risk of delayed anemia and subsequent top-up transfusions. However, other authors found that EPO may be less effective than expected. Due to the lack of evidence, routine use of EPO is currently not recommended. To determine a role for EPO in this group of patients, a well-designed randomized controlled clinical trial of sufficient sample size is required. Potentially, EPO stabilizes the hemoglobin levels of these infants and thus prevents top-up transfusions and extra admissions, creating a more stable and natural postnatal course for patients with HDN.

ELIGIBILITY:
Inclusion Criteria:

* all (near)-term neonates (gestational age ≥ 35 weeks) admitted to the Leiden University Medical Center (LUMC) with HDFN, treated with IUT.

Exclusion Criteria:

* none.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Number of top-up transfusions required per infant | First 3 months of life
  Number of top-up transfusions required per infant

SECONDARY OUTCOMES:
The percentage of infants requiring a top-up transfusion | First 3 months of life
  The percentage of infants requiring a top-up transfusion
Number of days of admission for top-up transfusions | First 3 months of life
  Number of days of admission for top-up transfusions
Occurrence of hypertension | 8 weeks (treatment course)
  The percentage of infants with a systolic blood pressure ≥ 2 SD above age adjusted mean systolic blood pressure during treatment
Occurrence of high ferritin levels | 8 weeks (treatment course)
  The percentage of infants with ferritin levels >200 μg/L during treatment

OTHER OUTCOMES:
Long-term neurodevelopmental outcome | 2 years of age
  Exploratory outcome; Long-term neurodevelopmental outcome at 2 years of age using the BSID-III test

CONTACTS AND LOCATIONS:
Overall Officials: Masja de Haas, MD PhD, Principal Investigator — Sanquin Research
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ree IMC, de Haas M, van Geloven N, Juul SE, de Winter D, Verweij EJT, Oepkes D, van der Bom JG, Lopriore E. Darbepoetin alfa to reduce transfusion episodes in infants with haemolytic disease of the fetus and newborn who are treated with intrauterine transfusions in the Netherlands: an open-label, single-centre, phase 2, randomised, controlled trial. Lancet Haematol. 2023 Dec;10(12):e976-e984. doi: 10.1016/S2352-3026(23)00285-5. PMID 38030319

DOCUMENTS (2):
  • Study Protocol (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT03104426/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03104426/SAP_001.pdf